CLINICAL TRIAL: NCT06571097
Title: Levofloxacin in the Treatment of Chronic Functional Constipation Associated With PIB Infection: A Multi-center, Exploratory Clinical Study
Brief Title: Levofloxacin in the Treatment of Chronic Functional Constipation Associated With PIB(Peristaltic Contraction-Inhibiting Bacterium) Infection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haifeng Lan (Other)
Responsible Party: Sponsor-Investigator, Haifeng Lan, student, Nanjing Medical University
Organization: Nanjing Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZQH-KYLL-24-20
Record Dates: First submitted 2024-08-06; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Constipation
Keywords: Levofloxacin; PIB; Peristaltic Contraction-Inhibiting Bacterium; constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Levofloxacin (Experimental): Levofloxacin: 0.5g(500mg)/day for 2 weeks
  Interventions: Drug: Levoﬂoxacin

INTERVENTIONS:
Drug: Levoﬂoxacin — 0.5g/day for 2 weeks

SUMMARY:
Constipation, a prevalent clinical condition, significantly impacts patients' quality of life, yet relevant clinical trial technical guidelines have yet to be issued domestically. This disease encompasses various classifications based on etiology, pathology, and pathophysiological characteristics. Slow transit constipation (STC), specifically, arises from colonic motility disorders and is recognized as a neuromuscular colonopathy. Currently, limited therapeutic options are available for patients with refractory STC, rendering it a common ailment associated with substantial disease burden and uncertain etiology. Consequently, identifying the cause and developing effective, targeted, and safe treatment strategies is of paramount importance.

Our research team has made a groundbreaking international discovery, revealing that STC is caused by infection with a novel Shigella-like bacterium, termed the peristaltic contraction-inhibiting bacterium (PIB), which secretes docosapentaenoic acid (DPA), an unsaturated fatty acid. The pathogenic mechanism involves inhibition of intestinal peristalsis, subsequently slowing colonic transit. Preliminary epidemiological studies confirm the exclusive presence of PIB in feces from patients with intractable constipation, whereas it is virtually absent in healthy individuals. Notably, consumption of high-dose DPA does not affect colonic transit or induce constipation; however, intracolonic administration does.

In response to PIB-induced STC, our team screened a range of antibiotics and identified two primary classes with potent antibacterial effects against PIB: fluoroquinolones and carbapenems. Both classes exhibit strong inhibitory activity against PIB, suggesting their potential use in chronic constipation treatment. Levofloxacin, a quinolone antibiotic, possesses broad-spectrum and potent antibacterial properties, effective in treating intestinal and urinary tract infections. Given that PIB has been confirmed as a novel Shigella-like species, and quinolones are established as the first-line antibiotics for Shigella infections, levofloxacin's efficacy against PIB was anticipated. Preliminary studies have validated levofloxacin's ability to inhibit PIB growth, thereby alleviating PIB-induced refractory constipation through sensitivity testing.

The primary objective of this study is to utilize levofloxacin to suppress PIB, thereby achieving the relief of chronic functional constipation.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to enter the trial.

1. Signed written informed consent;
2. Age 18-70;
3. Diagnosed chronic functional constipation according to Rome III or IV criteria, and infected with PIB;
4. Patients who have not taken other types of antibiotics in the past 1 month;
5. Bowel organic lesions (tumors and severe inflammatory lesions, etc.) were excluded by colonoscopy in the past 2 years.
6. The subjects could follow the follow-up plan, objectively describe the symptoms, and cooperate with the completion of the scale; 7）Agree to maintain similar diet and activity levels from the screening visit to the end of the study;

Exclusion Criteria:

Exclusion criteria: Subjects must exclude all of the following conditions to enter the study.

1. Pregnant and lactating women;
2. Patients with drug-induced constipation, including constipation induced by opioids and antidepressants;
3. During the study period, changes in lifestyle and dietary habits are not recommended in principle;
4. Patients with diseases that affect the conduct or results of the study, such as mental illness, serious cardiopulmonary, liver and kidney diseases, history of gastrointestinal surgery, epilepsy, etc.
5. Those who cannot take samples and complete inspection items as required;
6. Allergic to levofloxacin; 7）Other researchers found it inappropriate to participate in the project for clinical manifestations or diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Total effective rate of levofloxacin in the treatment of chronic functional constipation. | 6 months
  Obvious effect: no defecation difficulty, the number of spontaneous defecation ≥3 times/week (no effort and time consuming when defecating, no feeling of inadequate defecation, normal stool characteristics, etc.); Effective: the difficulty of defecation is improved than before, and the number of autonomous defecation is not less than 3 times/week (one of the time-consuming and laborious defecation or improper defecation or abnormal stool characteristics occurs during defecation);Ineffective: The difficulty of defecation is no better than before, and the number of spontaneous defecation is less than 3 times/week.Total effective rate = (significant efficiency + effective rate) Number of cases/total number of cases ×100%.

SECONDARY OUTCOMES:
PIB concentration (DPA content of docosapentaenoic acid) | 6 months
  PIB concentration ( DPA content in intestinal stool)
Proportion of patients with first defecation | 24-48 hours
  Proportion of patients with complete spontaneous defecation within 24-48 hours after receiving the first dose
Time of first defecation | 24-48 hours
  The time of patients with complete spontaneous defecation within 24-48 hours after receiving the first dose.
Number of frequency of use of rescue drugs and other Other defecation medications per week | 6 months
  Number of frequency of use of rescue drugs and other Other defecation medications per week
PAC-SYM | 6 months
  PAC-SYM（Patient Assessment of Constipation symptom）
PAC-QoL scale | 6 months
  PAC-Qol (Quality of life scale）
Bristol scale | 6 months
  Bristol (stool property)
The incidence of serious adverse events | 6 months
  intestinal obstruction, hematochezia, elevated indicators of serious infection, severe bloating, diarrhea, etc.
Patient satisfaction with treatment survey | 6 months
  Satisfaction degree of patients with levofloxacin treatment of constipation symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Levofloxacin in the Treatment of Chronic Functional Constipation Associated With PIB Infection: A Multi-center, Exploratory Clinical Study, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No